CLINICAL TRIAL: NCT02472938
Title: Phase IV, Interventional, multicenteR, Double-blind, Randomized, Placebo-controlled Study tO Explore the Onset of Efficacy on Magnetic Resonance Disease Activity of BG00012 (Dimethyl Fumarate) in Patients With relapsingremitTing Multiple Sclerosis
Brief Title: Study to Explore the Onset of Efficacy on Magnetic Resonance Disease Activity of BG00012 (Dimethyl Fumarate) in Patients With Relapsing remitTing Multiple Sclerosis
Acronym: PROMPT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Biogen (Industry)
Collaborators: GB Pharma Services & Consulting s.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIIT0115; ITA-BGT-14-10682 (Other: Biogen)
Record Dates: First submitted 2015-05-11; First posted 2015-06-16 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Relapsing remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BG00012 (Experimental): 120 mg capsule oral twice daily (BID) during the first week and 240 mg BID thereafter.
  Interventions: Drug: dimethyl fumarate
- Placebo (Placebo Comparator): Placebo capsules orally twice a day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: dimethyl fumarate — dimethyl fumarate 120 mg capsules
  Other Names: DMF; Tecfidera; BG00012
  Arms: BG00012
Other: Placebo — Placebo for BG00012
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the early efficacy of treatment with BG00012 (dimethyl fumarate) 240 mg twice daily (BID) in the brain of newly diagnosed and naive-to-treatment patients with relapsing-remitting multiple sclerosis (RRMS). The Secondary objectives are to establish the time course of the beneficial effect of BG00012 240 mg BID over 24 weeks and to evaluate the safety of BG00012.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with RRMS (McDonald criteria, 2010) who do not accept current injectable firstline DMTs.
* Multiple sclerosis (MS) onset within one year before enrolment
* ≥ 1 Gd+ lesions at a brain MRI scan performed within three months beforeenrolment.
* No previous disease modifying and/or immunosuppressive treatments for MS.
* Must have a baseline EDSS between 0.0 and 5.0, inclusive. · Women of childbearing potential (i.e. who are not post-menopausal for at least 1 year) and men must practice effective contraception (as defined by the Investigator) during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.

Exclusion Criteria:

* Primary progressive, secondary progressive, or progressive relapsing MS, as defined by Lublin and Reingold (Lublin and Reingold 1996)
* Previous disease modifying and/or immunosuppressive treatments for MS, including Tcell or T-cell receptor vaccination, any therapeutic monoclonal antibody, Mitoxantrone, Cyclophosphamide
* Previous treatment with Fumaderm®, dimethyl fumarate or other fumarates
* History of malignancy (except basal cell carcinoma that has been completely excised prior to study enrollment)
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity.Known allergy/hypersensitivity to Gadolinium.
* History of abnormal laboratory results indicative of any significant endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, renal, and/or other major disease that in the opinion of the Investigator would preclude participation in a clinical trial.
* History of or positive test result at screening for human immunodeficiency virus (HIV).Positive for hepatitis C antibody and/or positive for hepatitis B surface antigen (HBsAg) at screening.
* History of drug or alcohol abuse (as defined by the Investigator) within the 2 years prior to inclusion.
* An MS relapse that has occurred within the 30 days prior to inclusion (screening) AND/OR the subject has not stabilized from a previous relapse prior to inclusion.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Mean number of cumulative combined unique active (CUA) lesions (registered from week 4 to 24) | Week 24

SECONDARY OUTCOMES:
Mean number of CUA | at 4, 8, 12, 16, 20 and 24 weeks
Mean number of hypointense T1 lesions | at 24 weeks
New Gd+ lesions | at 4, 8, 12, 16, 20 and 24 weeks
New/enlarging T2 lesions | at 4, 8, 12, 16, 20 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen